CLINICAL TRIAL: NCT01109940
Title: An Open Label Non-randomized Extension Study to Evaluate the Safety and Tolerability of AIN457 (Anti Interleukin-17 Monoclonal Antibody) in Patients With Moderate to Severe Ankylosing Spondylitis
Brief Title: Safety and Tolerability of AIN457 in Adults (18-65 Years) With Moderate to Severe Ankylosing Spondylitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAIN457A2209E1; 2009-011591-30
Record Dates: First submitted 2010-04-22; First posted 2010-04-23 (Estimated); Results first posted 2021-06-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing spondylitis; IgG1K monoclonal antibody; Interleukin -17A neutralizing
MeSH Terms: conditions — Spondylitis, Ankylosing

ARMS (1):
- AIN457 (Experimental)
  Interventions: Biological: AIN457A

INTERVENTIONS:
Biological: AIN457A

SUMMARY:
This study is designed as an extension study to the proof-of-concept trial CAIN457A2209 in patients with moderate to severe ankylosing spondylitis and aims to provide continuous treatment with AIN457 for patients in the core trial, to obtain safety and tolerability information. The study will address the evaluation of efficacy following doses of Intravenous infusion (IV) of 3 mg/kg AIN457 given every 4 weeks over a period initially up to 6 months (Part 1) and based on the risk/benefit balance of AIN457 in ankylosing spondylitis a decision was taken to continue dosing for another 6 month period (Part 2).

ELIGIBILITY:
Inclusion Criteria:

* Patients who took part and completed in the core CAIN457A2209 study
* Patients who discontinued the core study due to unsatisfactory therapeutic effect at their Visit 14 (Week 16) or later could enter the extension study within 3 weeks of completing the study discontinuation visit of the core study, provided that at their discontinuation visit they fulfilled either one of the criteria below. Patients who did not enter the extension study within 3 weeks of completing the study discontinuation visit of the core study, were required to come for an additional baseline visit (Visit 17) and were required to fulfill either one of the criteria below:
* No improvement (compared with the core study baseline) in two out of the following four domains: patient global assessment, pain, BASFI and the mean of the two morning stiffness questions from the BASDAI. OR
* Deterioration (compared with the core study baseline) in one of the four domains (deterioration defined as >=20% worsening and an absolute worsening of >=1 unit)

Exclusion Criteria:

* Patients for whom continued treatment with AIN457 is not considered appropriate by the treating physician.
* Patients who were non-compliant or who demonstrated a major protocol deviation in the core CAIN457A2209 study.
* Patients who discontinued from the core CAIN457A2209 study before Visit 14 (Week 16), and patients who completed the core study
* Pregnant or lactating women
* Presence of active infection
* Positive PPD or HIV test in patients where repeated testing was deemed appropriate due to their risk profile

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (14):
- United States (8):
  - Novartis Investigative Site, Paradise Valley, Arizona
  - Novartis Investigative Site, Springfield, Illinois
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Duncansville, Pennsylvania
  - Novartis Investigative Site, Jackson, Tennessee
  - Novartis Investigative Site, Knoxville, Tennessee
  - Novartis Investigative Site, Benbrook, Texas
  - Novartis Investigative Site, Spokane, Washington
- Germany (4):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Herne
  - Novartis Investigative Site, München
- Novartis Investigative Site, Amsterdamn, DE, Netherlands
- Novartis Investigative Site, Newcastle upon Tyne, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 15 centers in four countries (Germany, Netherlands, United Kingdom, United States).
Pre-assignment Details: A total of 39 participants enrolled in the study of which 28 completed the study and 11 discontinued the study. Few participants were enrolled into the extension study (CAIN457A2209E1 [NCT01109940]) prior to completion of the core study (CAIN457A2209 [NCT00809159]).
Groups:
- Dose Group 1: Participants received 3 milligrams per kilogram (mg/kg) of intravenous (IV) secukinumab for every 4 weeks up to one year in the extension study (CAIN457A2209E1 [NCT01109940]) and who received secukinumab 2x10 mg/kg in the core study (CAIN457A2209 [NCT00809159]).
- Dose Group 2: Participants received 3 mg/kg of IV secukinumab for every 4 weeks up to one year in the extension study (CAIN457A2209E1 [NCT01109940]) and who received secukinumab 2x1.0 mg/kg in the core study (CAIN457A2209 [NCT00809159]).
- Dose Group 3: Participants received 3 mg/kg of IV secukinumab for every 4 weeks up to one year in the extension study (CAIN457A2209E1 [NCT01109940]) and who received secukinumab 2x0.1 mg/kg in the core study (CAIN457A2209 [NCT00809159]).
- Secukinumab/Placebo: Participants received 3 mg/kg of IV secukinumab for every 4 weeks up to one year in the extension study (CAIN457A2209E1 [NCT01109940]) and who received placebo in the core study (CAIN457A2209 [NCT00809159]).
Period: Overall Study
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Secukinumab/Placebo
Started | 21 | 8 | 7 | 3
Completed | 13 | 6 | 6 | 3
Not Completed | 8 | 2 | 1 | 0
Not completed — Administrative problems | 2 | 0 | 0 | 0
Not completed — Serious Adverse Event | 2 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Patient withdrew consent | 1 | 1 | 0 | 0
Not completed — Unsatisfactory therapeutic effect | 2 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Secukinumab/Placebo | Total
Number analyzed (Participants) | 21 | 8 | 7 | 3 | 39
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.5 (7.56) | 47.9 (11.27) | 45.9 (8.61) | 41.7 (11.59) | 42.5 (9.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 4 | 2 | 0 | 16
  Male | 11 | 4 | 5 | 3 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 18 | 8 | 6 | 3 | 35
  Other | 2 | 0 | 1 | 0 | 3
  Black | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reported Adverse Events (AE's)
Description: AEs are defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen.
Time Frame: From start of the study up to 64 weeks
Population: Safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Secukinumab/Placebo
Number analyzed (Participants) | 21 | 8 | 7 | 3
Participants | 21 | 6 | 6 | 3

2. Secondary Outcome: Number of Participants Reported Positive Antibodies for Secukinumab
Description: Immunogenicity (anti-drug antibodies) was assessed using an MSD bridging assay and a 3-tiered approach (screening, confirmation, titration).
Time Frame: Pre-dose, Week 0, 8, 24, 40 and Week 64
Population: Safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Secukinumab/Placebo
Number analyzed (Participants) | 21 | 8 | 7 | 3
Participants
  Week 0 | 0 | 0 | 0 | 0
  Week 8 | 0 | 0 | 0 | 0
  Week 24 | 0 | 0 | 0 | 0
  Week 40 | 0 | 0 | 0 | 0
  Week 64 | 0 | 0 | 0 | 0

3. Secondary Outcome: Total Interleukin (IL)- 17A Concentration in Blood at Steady-State
Description: Total serum IL17A was not measured due to assay limitations.
Time Frame: Pre-dose and at the end of infusion (up to 64 weeks)
Population: IL-17A measurements were planned for this study but could not be measured because the assay for total IL-17A, samples was not robust.
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Secukinumab/Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Maximum (Peak) Observed in Serum at Steady-State (Cmax,ss)
Description: Concentration of Secukinumab at the end of infusion (Cmax,ss) was reported.
Time Frame: At end of infusion (Week 64)
Population: All completed participants with quantifiable pharmacokinetics (PK) measurements and no major protocol deviations with impact on PK data were included in the PK analysis set. Here, the number of participants analyzed refer to the participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (μg/mL)
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Secukinumab/Placebo
Number analyzed (Participants) | 7 | 6 | 5 | 3
micrograms per milliliter (μg/mL) | 10.5 (3.03) | 10.6 (3.82) | 11.3 (4.81) | 17.1 (10.9)

5. Secondary Outcome: Minimum (Trough) Observed in Serum at Steady State (Cmin,ss)
Description: The concentration of secukinumab at pre-dose (Cmin,ss) in serum was reported.
Time Frame: Pre-dose (Week 0)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (μg/mL)
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Secukinumab/Placebo
Number analyzed (Participants) | 21 | 7 | 5 | 3
micrograms per milliliter (μg/mL) | 4.73 (10.1) | 15.0 (38.4) | 0.0428 (0.0586) | 27.1 (46.9)

ADVERSE EVENTS:
Time Frame: From Start of the Study up to 64 Weeks
Description: The analysis was performed on Safety analysis population (SAP) consisted of all participants who received at least one dose of study drug and had at least one valid post-baseline assessment.
Groups:
- Dose Group-1: Participants received 3 milligrams per kilogram (mg/kg) of intravenous (IV) secukinumab for every 4 weeks up to one year in the extension study (CAIN457A2209E1 [NCT01109940]) and who received secukinumab 2x10 mg/kg in the core study (CAIN457A2209 [NCT00809159]).
- Dose Group-2: Participants received 3 mg/kg of IV secukinumab for every 4 weeks up to one year in the extension study (CAIN457A2209E1 [NCT01109940]) and who received secukinumab 2x1.0 mg/kg in the core study (CAIN457A2209 [NCT00809159]).
- Dose Group-3: Participants received 3 mg/kg of IV secukinumab for every 4 weeks up to one year in the extension study (CAIN457A2209E1 [NCT01109940]) and who received secukinumab 2x0.1 mg/kg in the core study (CAIN457A2209 [NCT00809159]).
- Placebo/Secukinumab: Participants received 3 mg/kg of IV secukinumab for every 4 weeks up to one year in the extension study (CAIN457A2209E1 [NCT01109940]) and who received placebo in the core study (CAIN457A2209 [NCT00809159]).
Arm/Group | Dose Group-1 | Dose Group-2 | Dose Group-3 | Placebo/Secukinumab
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/8 | 0/7 | 0/3
Serious Adverse Events (participants affected / at risk) | 4/21 | 1/8 | 0/7 | 0/3
Other Adverse Events (participants affected / at risk) | 18/21 | 6/8 | 6/7 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Group-1 (N=21) | Dose Group-2 (N=8) | Dose Group-3 (N=7) | Placebo/Secukinumab (N=3)
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Group-1 (N=21) | Dose Group-2 (N=8) | Dose Group-3 (N=7) | Placebo/Secukinumab (N=3)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 2 | 1 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0
Iritis (Eye disorders) | 2 | 1 | 0 | 1
Uveitis (Eye disorders) | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Catheter site inflammation (General disorders) | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 3 | 2 | 0 | 1
Influenza like illness (General disorders) | 3 | 1 | 0 | 0
Oedema peripheral (General disorders) | 2 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Eye infection (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 0 | 0
Infected dermal cyst (Infections and infestations) | 0 | 1 | 1 | 0
Influenza (Infections and infestations) | 0 | 2 | 0 | 0
Nasopharyngitis (Infections and infestations) | 10 | 0 | 2 | 2
Paronychia (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Procedural headache (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Articular disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bone swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 2 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1
Mood swings (Psychiatric disorders) | 0 | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 1
Gynaecomastia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 1
Staphylococcal abscess (Infections and infestations) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No